CLINICAL TRIAL: NCT02878876
Title: Incidence of Lactose Intolerance Among Self-reported Lactose Intolerant People
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: a2 Milk Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 15-SC-11-A2-004
Record Dates: First submitted 2016-08-16; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Lactose Intolerance
MeSH Terms: conditions — Lactose Intolerance | interventions — Milk

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sequence A1-A2 (Experimental): Dietary Supplement: Oral consumption of milk with sequence A1-A2
  Interventions: Dietary Supplement: Oral consumption of milk with sequence A1-A2
- Sequence A2-A1 (Experimental): Dietary Supplement: Oral consumption of milk with sequence A2-A1
  Interventions: Dietary Supplement: Oral consumption of milk with sequence A2-A1

INTERVENTIONS:
Dietary Supplement: Oral consumption of milk with sequence A1-A2 — Oral consumption of 300 ml of milk containing both A1 and A2 type beta casein at 8:00 a.m. on Visit 1 (after 12-hour fasting) and 300 ml of milk containing only A2 type beta casein at 8:00 a.m. on Visit 2 (after 12-hour fasting).
  Arms: Sequence A1-A2
Dietary Supplement: Oral consumption of milk with sequence A2-A1 — Oral consumption of 300 ml of milk containing only A2 type beta casein at 8:00 a.m. on Visit 1 (after 12-hour fasting) and 300 ml of milk containing both A1 and A2 type beta casein at 8:00 a.m. on Visit 2 (after 12-hour fasting).
  Arms: Sequence A2-A1

SUMMARY:
This is a 3-sites, double-blinded, randomized, 2X2 cross-over study aiming to compare effects of milk containing only A2 type beta casein versus milk containing both A1 and A2 beta casein proteins on the gastrointestinal symptoms for the health people who self-reported to be lactose intolerant.

DETAILED DESCRIPTION:
Study sites: Shanghai, Guangzhou, Beijing

Eligible subjects were enrolled in the study and randomized into one of the 2 study arms:

Sequence A1-A2: Oral consumption of milk containing both A1 and A2 type beta casein at Visit 1 and milk containing only A2 type beta casein at Visit 2; Sequence A2-A1: Oral consumption of milk containing only A2 type beta casein at Visit 1 and milk containing both A1 and A2 type beta casein at Visit 2.

Washout period: 2 weeks between Visit 1 and Visit 2

ELIGIBILITY:
Inclusion Criteria:

* 20~50 years old male or female subjects;
* Non-regular milk drinker with self-reported intolerance to commercial milk;
* Suffered from mild to moderate digestive discomfort after milk consumption;
* Have normal electrocardiograms (ECG) and blood pressure during quiet respiration;
* Agree not to take any medication, supplements, nutrition or other dairy products including acidophilus milk;
* Be willing to comply with all the requirements and procedures of the study;
* Agree to sign the informed consent form;
* Agree not to enroll in another interventional clinical research study while participating in this study;
* Fully understand the nature, objective, benefit and the potential risks and side effects of the study.

Exclusion Criteria:

* Female on pregnant or feeding；
* Have known dairy allergy;
* Have severe response to milk intolerance;
* Have history of faecal impaction;
* Trying to lose weight by following a diet or exercise regimen designed for weight loss, or taking any drug influencing appetite and any drug for weight loss for the last three months ;
* Have participated in similar dairy or probiotics-containing product's clinical trials within 3 months before the screening;
* Currently taking medicines for cardiovascular or metabolic disease;
* Have history of or be diagnosed of any of the following diseases that may affect the study results: gastrointestinal disorders, hepatopathy, nephropathy, endocrine disease, blood disorders, respiratory and cardiovascular diseases;
* Current or previous alcohol abuser, currently taking or took illicit drugs, substance or OTC prescription drugs in regular frequency which may affect gastrointestinal disorders and study result;
* Currently suffering from any gastrointestinal disorders or gastrointestinal disease, including but not limited to: irritable bowel syndrome, colitis, ulcerative colitis, celiac disease, irritable bowel syndrome(IBS);
* Had hospitalizations within 3 months before screening;
* Currently drug frequency user of that may affect the gastrointestinal function or immune system. As judged by investigator.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal Symptom VAS scores at 3 hours | Three hours after product intervention at each of Visit 1 and Visit 2
  Gastrointestinal symptoms were self-measured by study subjects on a scale from 0 (not at all) to 9 (severe) at 3 hours after product consumption at Visit 1 and Visit 2. Data was analyzed as a repeated measures design using a mixed effects ANOVA with symptom VAS scores at 3-hour as outcome, study product (A1 or A2) and study visit (1 or 2) as fixed effects, and a random subject effect nested within the sequence of study treatment (A1-A2 or A2-A1) , and adjusted for baseline symptom scores. Type III tests of fixed effects were used for testing the effect of study products. Contrast tests were generated to compare means for each product.

SECONDARY OUTCOMES:
The percentage of improvement in gastrointestinal symptoms after drinking A2 versus A1 | 1 hour and 3 hours after product intervention
  The improvement in gastrointestinal symptoms after drinking A2 versus A1 were classified into 4 mutually exclusive categories according to the following definition:
  * No symptom: have no gastrointestinal symptoms after drinking product A2 while having symptoms after drinking product A1.
  * Significant improvement: still have gastrointestinal symptom after drinking product A2, the reduction of symptom scores >3
  * Slight improvement: still have gastrointestinal symptom after drinking product A2, 1<=reduction of symptom scores<=3
  * No difference (not improved or worsen): reduction of symptom scores<=0
  The frequency and percentage in each category of improvement for each single gastrointestinal symptom, as well as that for all symptoms, are summarized.
Urinary galactose concentration | baseline and 3 hours after product intervention of each of Visit 1 and Visit 2
  Urinary galactose (U-gal) concentration was measured at baseline and 3-hour of each of Visit 1 and Visit 2. Data was analyzed as a repeated measures design using a mixed effects ANOVA with fixed effects of study product (A1 or A2) and study visit (1 or 2) and a random subject effect nested within the sequence of study treatment (A1-A2 or A2-A1) , and adjusted for baseline symptom scores. Type III tests of fixed effects were used for testing the effect of study products. Contrast tests were generated to compare means for each product.
  The U-gal measurements over the whole study period (both Visit 1 and Visit 2) for all subjects were also summarized by study product. Product difference was evaluated using one-way ANOVA.
Gastrointestinal Symptom VAS scores at 1 hour | One hour after product intervention at each of Visit 1 and Visit 2
  Gastrointestinal symptoms were self-measured by study subjects on a scale from 0 (not at all) to 9 (severe) at 1 hour after product consumption at Visit 1 and Visit 2. Data was analyzed as a repeated measures design using a mixed effects ANOVA with symptom VAS scores at 1-hour as outcome, study product (A1 or A2) and study visit (1 or 2) as fixed effects, and a random subject effect nested within the sequence of study treatment (A1-A2 or A2-A1) , and adjusted for baseline symptom scores. Type III tests of fixed effects were used for testing the effect of study products. Contrast tests were generated to compare means for each product.
Change of urinary galactose concentration from baseline at 3 hours <0.27 mmol/L (Yes/No) | 3 hours after product intervention of each of Visit 1 and Visit 2
  Based on the results of urinary galactose test, subjects were classified as lactose malabsorbers if they had an increase in urinary galactose concentration of <0.27 mmol/L at 3 hours after oral consumption of 15g lactose (corresponding to 300 ml of product A1). And those with an increase in urinary galactose concentration of ≥0.27 mmol/L at 3-hour were classified as lactose absorbers.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Clarke, PhD, Study Director — a2 Milk Company Ltd.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He M, Sun J, Jiang ZQ, Yang YX. Effects of cow's milk beta-casein variants on symptoms of milk intolerance in Chinese adults: a multicentre, randomised controlled study. Nutr J. 2017 Oct 25;16(1):72. doi: 10.1186/s12937-017-0275-0. PMID 29070042